CLINICAL TRIAL: NCT00407511
Title: A Prospective, Open Label, Multi-Center, Study Of Pregabalin In The Treatment Of Neuropathic Pain Associated With Diabetic Peripheral Neuropathy, Postherpetic Neuralgia, HIV-Related Peripheral Neuropathic Pain And Chemotherapy Induced Peripheral Neuropathic Pain
Brief Title: Pregabalin Treatment Of Peripheral Neuropathic Pain Associated With Diabetic Peripheral NeP (DPN), Postherpetic Neuralgia (PHN), HIV-related NeP (HIV), and Chemotherapy Induced NeP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A0081097
Record Dates: First submitted 2006-12-01; First posted 2006-12-05 (Estimated); Results first posted 2009-08-19 (Estimated); Last update posted 2021-02-09 (Actual); Status verified 2009-10

CONDITIONS: Diabetic Peripheral Neuropathic Pain (DPN); Postherpetic Neuralgia (PHN); HIV-related Neuropathic Pain (HIV); Chemotherapy Induced Neuropathic Pain
MeSH Terms: conditions — Neuralgia, Postherpetic | interventions — Pregabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pregabalin (Experimental)
  Interventions: Drug: Pregabalin

INTERVENTIONS:
Drug: Pregabalin — Pregabalin will be administered orally, twice a day for 12 weeks, including 4-week dose adjustment phase followed by 8-week maintenance phase. The minimum allowable pregabalin dose during the trial will be 75 mg BID (150 mg/day) and the maximum allowable dose will be 300 mg BID (600 mg/day).

SUMMARY:
Management of neuropathic pain associated with diabetic peripheral neuropathy, post-herpetic neuralgia, human immunodeficiency virus-related peripheral neuropathy, and chemotherapy induced peripheral neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are diagnosed with neuropathic pain associated with diabetic peripheral neuropathy, post-herpetic neuralgia, human immunodeficiency virus related peripheral neuropathy, and chemotherapy induced peripheral neuropathy.

Exclusion Criteria:

* Severe Pain associated with conditions other than Diabetic Peripheral Neuropathy, Post-Herpetic Neuralgia, Human Immunodeficiency virus related peripheral neuropathy, and chemotherapy induced peripheral neuropathy that may confound assessment or self evaluation of the neuropathic pain.
* Skin Condition in the affected dermatome that (in the judgment of the investigator) could alter sensation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2007-01; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (10):
- Pfizer Investigational Site, Bogota, Cundinamarca, Colombia
- Pfizer Investigational Site, Quito, Pichincha, Ecuador
- Mexico (6):
  - Pfizer Investigational Site, Tijuana, B. C.
  - Pfizer Investigational Site, Mexicali, B.C.
  - Pfizer Investigational Site, Acapulco de Juárez, Guerrero
  - Pfizer Investigational Site, Mexico City, Mexico City
  - Pfizer Investigational Site, México, Monterrey, NL
  - Pfizer Investigational Site, Mérida, Yucatán
- Pfizer Investigational Site, Lima, Peru
- Pfizer Investigational Site, Caracas, Distrito Federal, Venezuela

REFERENCES:
- [Derived] Xochilcal-Morales M, Castro EM, Guajardo-Rosas J, Obregon TN, Acevedo JC, Chucan JM, Plancarte-Sanchez R, Davila G, Wajsbrot D, Guerrero M, Vinueza R. A prospective, open-label, multicentre study of pregabalin in the treatment of neuropathic pain in Latin America. Int J Clin Pract. 2010 Aug;64(9):1301-9. doi: 10.1111/j.1742-1241.2010.02389.x. Epub 2010 May 10. PMID 20487048
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081097&StudyName=Pregabalin%20Treatment%20Of%20Peripheral%20Neuropathic%20Pain%20Associated%20With%20Post-Herpetic%2C%20%28HIV%2CChemotherapy%29%20Diabetic%20Induced

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at 13 medical centers in Latin America and participated between January 2007 and July 2008.
Pre-assignment Details: 160 subjects were screened and evaluated for inclusion/exclusion criteria; 121 were assigned to open-label treatment.
Groups:
- Pregabalin: Dose adjustment phase: Week 1: 75mg BID (150 mg/day) all subjects; Week 2 through Week 4: subjects were assessed on a weekly basis for dose adjustment from 75 mg BID (150 mg/day) to 150 mg BID (300 mg/day), and to 300 mg BID (600 mg/day) if needed based on pain relief and tolerability. 8 week dose maintenance phase (Week 5 to Week 12): subjects continued with their final pregabalin dosage: 75mg BID (150 mg/day) to 300 mg BID (600 mg/day) based on individual pain response and tolerability.
Period: Overall Study
Arm/Group | Pregabalin
Started | 121
Completed | 99
Not Completed | 22
Not completed — Adverse Event | 9
Not completed — Lost to Follow-up | 4
Not completed — Other | 5
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Arm/Group | Pregabalin
Number analyzed (Participants) | 121
Age, Customized [Number; unit: participants]
  Between 18 to 44 years | 15
  Between 45 to 64 years | 76
  >= 65 years | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83
  Male | 38

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to End of Treatment (EOT) in Weekly Mean Pain Score on the Daily Pain Rating Scale (DPRS)
Description: 11 point Likert scale: range 0 to 10 (no pain to worst possible pain) over past 24 hours. Baseline score = mean score of preceding 7 days (including Visit 2). Final end of treatment (EOT) pain score = mean pain score from last 7 post-Baseline days preceding Visit 8 (Week 12) or last 7 days on study drug for those who did not complete the study. Change = mean at EOT minus mean at Baseline.
Time Frame: Baseline, End of Treatment
Population: Full Analysis Set (FAS): patients who took at least one dose of study medication, had a baseline value, and had at least one post-baseline measurement; Last Observation Carried Forward (LOCF).
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | Pregabalin
Number analyzed (Participants) | 120
scores on scale | -3.8 (2.5)
Statistical Analysis 1: Comparison: Pregabalin; End of treatment/last observation carried forward (EOT/LOCF): value consists of the mean of the last 7 post-baseline visits scores. Mean change: the arithmetic mean change and p-value from the single sample t-test. If < = 7 and > = 4 post-baseline scores were available, the mean pain score was computed using the available scores. The mean was not calculated if there were less than 4 post-baseline scores prior to study termination; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

2. Secondary Outcome: Change From Baseline in Mean Pain Score on the Daily Pain Rating Scale (DPRS)
Description: 11 point Likert scale; range: 0 to 10 (no pain to worst possible pain) over past 24 hours. Baseline score = mean score of preceding 7 days (including Visit 2). Weekly pain score = mean pain score from last 7 post-Baseline days preceding observation visit or last 7 days on study drug for early termination. Change = mean at observation minus mean at Baseline.
Time Frame: Week 4, Week 8, Week 12
Population: Full Analysis Set (FAS).
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | Pregabalin
Number analyzed (Participants) | 120
scores on scale
  Week 4 (n=110) | -3.2 (1.9)
  Week 8 (n=100) | -3.9 (2.3)
  Week 12 (n=96) | -4.2 (2.4)
Statistical Analysis 1: Comparison: Pregabalin; Week 4; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -3.2, 95% CI [-3.6 to -2.8], Standard Error of Mean 0.2 — Parameter estimate: Mean Difference (Final Values) = least squares mean
Statistical Analysis 2: Comparison: Pregabalin; Week 8; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -3.9, 95% CI [-4.3 to -3.5], Standard Error of Mean 0.2 — Parameter estimate: Mean Difference (Final Values) = least squares mean
Statistical Analysis 3: Comparison: Pregabalin; Week 12; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -4.1, 95% CI [-4.5 to -3.7], Standard Error of Mean 0.2 — Parameter estimate: Mean Difference (Final Values) = least squares mean

3. Secondary Outcome: Change From Baseline (BL) in Modified Brief Pain Inventory-Short Form (m-BPI-sf): Pain Severity Index Scores
Description: Self-administered questionnaire: change from Baseline in mean pain severity index over past 24 hours; 11-point numeric rating scale ranging from 0 (no pain) to 10 (worst pain possible). Pain severity index is the mean of item scores 2, 3, and 4 (pain right now, worst pain, and average pain level). Change = mean score at observation minus mean score at Baseline.
Time Frame: Baseline, Week 8, Week 12, EOT/LOCF
Population: Full Analysis Set (FAS); End of Treatment/Last Observation Carried Forward (EOT/LOCF): last post-baseline assessment.
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | Pregabalin
Number analyzed (Participants) | 120
scores on scale
  Week 8 (n=102) | -4.2 (2.6)
  Week 12 (n=98) | -4.7 (2.6)
  EOT/LOCF (n=102) | -4.6 (2.6)
Statistical Analysis 1: Comparison: Pregabalin; Week 8, FAS. Week 8: subjects were only included if their visit fell within the computed week (49 to 63 days); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -4.2, 95% CI [-4.7 to -3.7], Standard Error of Mean 0.2 — Parameter estimate: Mean Difference (Final Values) = least squares mean
Statistical Analysis 2: Comparison: Pregabalin; Week 12: subjects were only included if their visit fell within the computed week (>= 78 days); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -4.6, 95% CI [-5.1 to -4.1], Standard Error of Mean 0.2 — Parameter estimate: Mean Difference (Final Values) = least squares mean
Statistical Analysis 3: Comparison: Pregabalin; EOT/LOCF: last post-baseline value; mean change from Baseline was the arthmetic mean change and the p-value was from the single-sample t-test; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

4. Secondary Outcome: Change From Baseline in Modified Brief Pain Inventory-Short Form (m-BPI-sf): Pain Interference Index Scores
Description: Self-administered questionnaire: change from Baseline in mean pain interference with functional activities (general activity, mood, walking ability, relations with other people, sleep, normal work, and enjoyment of life) in past 24 hours. 11-point scale from 0 (does not interfere) to 10 (completely interferes). Change = observation mean minus Baseline mean.
Time Frame: Baseline, Week 8, Week 12, End of Treatment/Last Observation Carried Forward (EOT/LOCF)
Population: Full Analysis Set (FAS); End of Treatment/Last Observation Carried Forward (EOT/LOCF): last post-baseline assessment.
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | Pregabalin
Number analyzed (Participants) | 120
scores on scale
  Week 8 (n=102) | -3.8 (2.7)
  Week 12 (n=98) | -4.2 (2.6)
  EOT/LOCF (n=102) | -4.0 (2.6)
Statistical Analysis 1: Comparison: Pregabalin; Week 8: subjects were only included if their visit fell within the computed week (Day 49 to 63); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -3.8, 95% CI [-4.2 to -3.4], Standard Error of Mean 0.2 — Parameter estimate: Mean Difference (Final Values) = least squares mean
Statistical Analysis 2: Comparison: Pregabalin; Week 12: subjects were only included if their visit fell within the computed week (>= Day 78); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -4.1, 95% CI [-4.5 to -3.7], Standard Error of Mean 0.2 — Parameter estimate: Mean Difference (Final Values) = least squares mean
Statistical Analysis 3: Comparison: Pregabalin; [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

5. Secondary Outcome: Pain Treatment Satisfaction Scale (PTSS): Impact of Current Pain Medication
Description: Impact of current pain medication response scale: 0 (worst possible response) to 100 (best possible response). Score=[(5-mean of non-missing items)*100]/4.
Time Frame: Baseline, Week 8, Week 12, EOT/LOCF
Population: Full Analysis Set (FAS); End of Treatment/Last Observation Carried Forward (EOT/LOCF): last post-baseline assessment. Subjects were only included in the Week 8 analysis if their visit fell between Days 49 and 63, and were only included in the Week 12 analysis if their visit was after Day 78.
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | Pregabalin
Number analyzed (Participants) | 105
scores on scale
  Baseline (n=78) | 62.34 (29.99)
  Week 8 (n=100) | 90.38 (16.17)
  Week 12 (n=97) | 91.66 (13.83)
  EOT/LOCF (n=105) | 91.40 (14.95)

6. Secondary Outcome: Pain Treatment Satisfaction Scale (PTSS): Satisfaction With Current Pain Medication
Description: Satisfaction with current pain medication response scale: 0 (worst possible response) to 100 (best possible response). Score=[(5-mean of non-missing items)*100]/4.
Time Frame: Baseline, Week 8, Week 12, EOT/LOCF
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | Pregabalin
Number analyzed (Participants) | 105
scores on scale
  Baseline (n=78) | 52.56 (24.68)
  Week 8 (n=100) | 85.92 (16.96)
  Week 12 (n=97) | 88.56 (13.87)
  EOT/LOCF (n=105) | 88.08 (14.72)

7. Secondary Outcome: Change From Baseline in Visual Analogue Scale for Pain (VAS-pain)
Description: 100 mm line (Visual Analog Scale) marked by subject; Intensity of pain range (over past week): 0 = no pain to 100 = worst possible pain. Change = observation mean minus Baseline mean.
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4, Week 8, Week 12, EOT/LOCF
Population: Full Analysis Set (FAS); End of Treatment/Last Observation Carried Forward (EOT/LOCF): last post-baseline assessment.
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | Pregabalin
Number analyzed (Participants) | 120
scores on scale
  Week 1 (n = 120) | -18.8 (21.9)
  Week 2 (n = 116) | -28.5 (24.1)
  Week 3 (n = 116) | -34.9 (25.8)
  Week 4 (n = 109) | -41.0 (24.6)
  Week 8 (n = 102) | -46.6 (26.2)
  Week 12 (n = 98) | -49.0 (26.6)
  EOT/LOCF (n = 120) | -45.9 (28.8)
Statistical Analysis 1: Comparison: Pregabalin; Week 1: LS mean, p-value, and confidence interval are based on a repeated measures mixed effect model with baseline value, center, and week as fixed effects; subject was included as a random effect. Subjects were only included in the Week 1 assessment if their visit fell within Days 4 to 10; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -18.1, 95% CI [-22.3 to -14.0], Standard Error of Mean 2.1 — Parameter estimate: Mean Difference (Final Values) = least squares mean
Statistical Analysis 2: Comparison: Pregabalin; Week 2: LS mean, p-value, and confidence interval are based on a repeated measures mixed effect model with baseline value, center, and week as fixed effects; subject was included as a random effect. Subjects were only included in the Week 2 assessment if their visit fell within Days 11 to 17; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Median Difference (Final Values) = -28.2, 95% CI [-32.4 to -24.0], Standard Error of Mean 2.1 — Parameter estimate: Mean Difference (Final Values) = least squares mean
Statistical Analysis 3: Comparison: Pregabalin; Week 3: LS mean, p-value, and confidence interval are based on a repeated measures mixed effect model with baseline value, center, and week as fixed effects; subject was included as a random effect. Subjects were only included in the Week 3 assessment if their visit fell within Days 18 to 24; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -34.3, 95% CI [-38.5 to -30.0], Standard Error of Mean 2.1 — Parameter estimate: Mean Difference (Final Values) = least squares mean
Statistical Analysis 4: Comparison: Pregabalin; Week 4: LS mean, p-value, and confidence interval are based on a repeated measures mixed effect model with baseline value, center, and week as fixed effects; subject was included as a random effect. Subjects were only included in the Week 4 assessment if their visit fell within days 25 to 35; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -40.9, 95% CI [-45.2 to -36.7], Standard Error of Mean 2.2 — Parameter estimate: Mean Difference (Final Values) = least squares mean
Statistical Analysis 5: Comparison: Pregabalin; Week 8: LS mean, p-value, and confidence interval are based on a repeated measures mixed effect model with baseline value, center, and week as fixed effects; subject was included as a random effect. Subjects were only included in the Week 8 assessment if their visit fell within Days 49 to 63; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -45.8, 95% CI [-50.2 to -41.4], Standard Error of Mean 2.2 — Parameter estimate: Mean Difference (Final Values) = least squares mean
Statistical Analysis 6: Comparison: Pregabalin; Week 12: LS mean, p-value, and confidence interval are based on a repeated measures mixed effect model with baseline value, center, and week as fixed effects; subject was included as a random effect. Subjects were only included in the Week 12 assessment if their visit fell >= Day 78; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -48.4, 95% CI [-52.8 to -44.0], Standard Error of Mean 2.2 — Parameter estimate: Mean Difference (Final Values) = least squares mean
Statistical Analysis 7: Comparison: Pregabalin; EOT/LOCF: last post-baseline assessment. Mean change is the arithmetic mean change; p-value is from a single-sample t-test; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

8. Secondary Outcome: Change From Baseline in Global Anxiety Visual Analogue Scale (GA-VAS)
Description: 100-mm line (Visual Analog Scale) marked by the subject to measure their degree of anxiety over past 24 hours. Range: 0 = not at all anxious to 100 = extremely anxious. Change = mean score at observation minus mean score at Baseline.
Time Frame: Baseline, Week 8, Week 12, EOT/LOCF
Population: Full Analysis Set (FAS); End of Treatment/Last Observation Carried Forward (EOT/LOCF): last post-baseline assessment.
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | Pregabalin
Number analyzed (Participants) | 118
scores on scale
  Week 8 (n=99) | -39.2 (29.6)
  Week 12 (n=97) | -41.4 (32.9)
  EOT/LOCF (n=101) | -40.5 (33.1)
Statistical Analysis 1: Comparison: Pregabalin; Week 8: LS mean, p-value, and confidence interval are based on a repeated measures effect model with baseline value, center, and week as fixed effects; subjects were included as a random effect. Subjects were included in the Week 8 assessment only if their visit fell within Days 49 and 63; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -38.7, 95% CI [-43.4 to -33.9], Standard Error of Mean 2.4 — Parameter estimate: Mean Difference (Final Values) = least squares mean
Statistical Analysis 2: Comparison: Pregabalin; Week 12: LS mean, p-value, and confidence interval are based on a repeated measures effect model with baseline value, center, and week as fixed effects; subjects were included as a random effect. Subjects were included in the Week 12 assessment only if their visit fell >=Day 78; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -40.7, 95% CI [-45.5 to -35.9], Standard Error of Mean 2.4 — Parameter estimate: Mean Difference (Final Values) = least squares mean
Statistical Analysis 3: Comparison: Pregabalin; EOT/LOCF: last post-baseline assessment. Mean change= arithmetic mean change; p-value is from a single-sample t-test; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

9. Secondary Outcome: Change From Baseline in Mean Daily Sleep Interference Score (DSIS)
Description: Daily sleep interference measured on an 11-point Likert scale. Range: 0 (pain did not interfere with sleep) to 10 (pain completely interfered with sleep). Change = mean at observation minus mean at Baseline. Evaluations recorded in patient's daily sleep diaries.
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, Week 8, Week 9, Week 10, Week 11, Week 12, EOT/LOCF
Population: Full Analysis Set (FAS); End of Treatment/Last Observation Carried Forward (EOT/LOCF): last post-baseline assessment.
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | Pregabalin
Number analyzed (Participants) | 120
scores on scale
  Week 1 (n=120) | -1.0 (1.5)
  Week 2 (n=118) | -1.8 (2.0)
  Week 3 (n=114) | -2.5 (2.2)
  Week 4 (n=110) | -2.8 (2.3)
  Week 5 (n=104 | -3.0 (2.3)
  Week 6 (n=103) | -3.1 (2.5)
  Week 7 (n=100) | -3.3 (2.5)
  Week 8 (n=100) | -3.4 (2.5)
  Week 9 (n=97) | -3.5 (2.6)
  Week 10 (n=99) | -3.5 (2.7)
  Week 11 (n=98) | -3.5 (2.6)
  Week 12 (n=96) | -3.4 (2.7)
  EOT/LOCF (n=120) | -3.1 (2.7)
Statistical Analysis 1: Comparison: Pregabalin; Week 1: LS mean, p-value, and confidence interval are based on repeated measures mixed effect model with baseline value, pooled center, and weeks 1, 4, 8 and 12 as fixed effects; subjects were included as a random effect; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -1.0, 95% CI [-1.4 to -0.7], Standard Error of Mean 0.2 — Parameter estimate: Mean Difference (Final Values) = least squares mean
Statistical Analysis 2: Comparison: Pregabalin; Week 2: LS mean, p-value, and confidence interval are based on repeated measures mixed effect model with baseline value, pooled center, and weeks 1, 4, 8 and 12 as fixed effects; subjects were included as a random effect; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -1.8, 95% CI [-2.2 to -1.5], Standard Error of Mean 0.2 — Parameter estimate: Mean Difference (Final Values) = least squares mean
Statistical Analysis 3: Comparison: Pregabalin; Week 3: LS mean, p-value, and confidence interval are based on repeated measures mixed effect model with baseline value, pooled center, and weeks 1, 4, 8 and 12 as fixed effects; subjects were included as a random effect; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -2.5, 95% CI [-2.9 to -2.2], Standard Error of Mean 0.2 — Parameter estimate: Mean Difference (Final Values) = least squares mean
Statistical Analysis 4: Comparison: Pregabalin; Week 4: LS mean, p-value, and confidence interval are based on repeated measures mixed effect model with baseline value, pooled center, and weeks 1, 4, 8 and 12 as fixed effects; subjects were included as a random effect; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -2.8, 95% CI [-3.2 to -2.5], Standard Error of Mean 0.2 — Parameter estimate: Mean Difference (Final Values) = least squares mean
Statistical Analysis 5: Comparison: Pregabalin; Week 5: LS mean, p-value, and confidence interval are based on repeated measures mixed effect model with baseline value, pooled center, and weeks 1, 4, 8 and 12 as fixed effects; subjects were included as a random effect; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -2.9, 95% CI [-3.3 to -2.6], Standard Error of Mean 0.2 — Parameter estimate: Mean Difference (Final Values) = least squares mean
Statistical Analysis 6: Comparison: Pregabalin; Week 6: LS mean, p-value, and confidence interval are based on repeated measures mixed effect model with baseline value, pooled center, and weeks 1, 4, 8 and 12 as fixed effects; subjects were included as a random effect; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -3.0, 95% CI [-3.4 to -2.6], Standard Error of Mean 0.2 — Parameter estimate: Mean Difference (Final Values) = least squares mean
Statistical Analysis 7: Comparison: Pregabalin; Week 7: LS mean, p-value, and confidence interval are based on repeated measures mixed effect model with baseline value, pooled center, and weeks 1, 4, 8 and 12 as fixed effects; subjects were included as a random effect; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -3.1, 95% CI [-3.5 to -2.8], Standard Error of Mean 0.2 — Parameter estimate: Mean Difference (Final Values) = least squares mean
Statistical Analysis 8: Comparison: Pregabalin; Week 8: LS mean, p-value, and confidence interval are based on repeated measures mixed effect model with baseline value, pooled center, and weeks 1, 4, 8 and 12 as fixed effects; subjects were included as a random effect; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -3.2, 95% CI [-3.6 to -2.8], Standard Error of Mean 0.2 — Parameter estimate: Mean Difference (Final Values) = least squares mean
Statistical Analysis 9: Comparison: Pregabalin; Week 9: LS mean, p-value, and confidence interval are based on repeated measures mixed effect model with baseline value, pooled center, and weeks 1, 4, 8 and 12 as fixed effects; subjects were included as a random effect; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -3.3, 95% CI [-3.7 to -2.9], Standard Error of Mean 0.2 — Parameter estimate: Mean Difference (Final Values) = least squares mean
Statistical Analysis 10: Comparison: Pregabalin; Week 10: LS mean, p-value, and confidence interval are based on repeated measures mixed effect model with baseline value, pooled center, and weeks 1, 4, 8 and 12 as fixed effects; subjects were included as a random effect; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -3.4, 95% CI [-3.7 to -3.0], Standard Error of Mean 0.2 — Parameter estimate: Mean Difference (Final Values) = least squares mean
Statistical Analysis 11: Comparison: Pregabalin; Visit 11: LS mean, p-value, and confidence interval are based on repeated measures mixed effect model with baseline value, pooled center, and weeks 1, 4, 8 and 12 as fixed effects; subjects were included as a random effect; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -3.4, 95% CI [-3.8 to -3.0], Standard Error of Mean 0.2 — Parameter estimate: Mean Difference (Final Values) = least squares mean
Statistical Analysis 12: Comparison: Pregabalin; Week 12: LS mean, p-value, and confidence interval are based on repeated measures mixed effect model with baseline value, pooled center, and weeks 1, 4, 8 and 12 as fixed effects; subjects were included as a random effect; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -3.4, 95% CI [-3.7 to -3.0], Standard Error of Mean 0.2 — Parameter estimate: Mean Difference (Final Values) = least squares mean
Statistical Analysis 13: Comparison: Pregabalin; EOT/LOCF value consists of the mean of the last 7 post-baseline sleep scores; mean change = arithmetic mean change; p-value: from single sample t-test; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

10. Secondary Outcome: Patient Global Impression of Change (PGIC)
Description: 7-point participant rating scale for change observed in their overall status since beginning of study medication. Range: 1 (very much improved) to 7 (very much worse)
Time Frame: End of Treatment/ Last Observation Carried Forward (Week 12 or last post-baseline assessment)
Population: Full Analysis Set (FAS)
Measure: Number; unit: participants
Arm/Group | Pregabalin
Number analyzed (Participants) | 103
participants
  Very much improved | 37
  Much improved | 53
  Minimally improved | 12
  No change | 1
  Minimally worse | 0
  Much worse | 0
  Very much worse | 0

11. Secondary Outcome: Clinical Global Impression of Change (CGIC)
Description: 7-point investigator rating scale of change in participant's status since beginning study medication. Range: 1 (very much improved) to 7 (very much worse).
Time Frame: End of Treatment/ Last Observation Carried Forward (Week 12 or last post-baseline assessment)
Population: Full Analysis Set (FAS)
Measure: Number; unit: participants
Arm/Group | Pregabalin
Number analyzed (Participants) | 103
participants
  Very much improved | 41
  Much improved | 55
  Minimally improved | 5
  No change | 2
  Minimally worse | 0
  Much Worse | 0
  Very much worse | 0

ADVERSE EVENTS:
Arm/Group | Pregabalin
Serious Adverse Events (participants affected / at risk) | 4
Other Adverse Events (participants affected / at risk) | 69
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Pregabalin
Cardiac failure (Cardiac disorders) | 1/121
Pericarditis (Cardiac disorders) | 1/121
Vitreous haemorrhage (Eye disorders) | 1/121
Generalized oedema (General disorders) | 1/121
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 1/121
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/121
Headache (Nervous system disorders) | 1/121
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Pregabalin
Dry mouth (Gastrointestinal disorders) | 8/121
Nausea (Gastrointestinal disorders) | 6/121
Oedema (General disorders) | 7/121
Oedema peripheral (General disorders) | 14/121
Weight increased (Investigations) | 15/121
Increased appetite (Metabolism and nutrition disorders) | 7/121
Dizziness (Nervous system disorders) | 25/121
Headache (Nervous system disorders) | 8/121
Somnolence (Nervous system disorders) | 38/121

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.